CLINICAL TRIAL: NCT03342560
Title: Beyond Confounders: Addressing Source of Measurement Variability and Error in Shear Wave Elastography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Canon Medical Systems, USA (Industry); Siemens Medical Solutions (Industry); Radiological Society of North America (Other)
Responsible Party: Principal Investigator, Anthony Samir, Service Chief,Body Ultrasound Department of Radiology, Assistant Professor at Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017P000940
Record Dates: First submitted 2017-11-06; First posted 2017-11-17 (Actual); Results first posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Liver Fibrosis; Liver Diseases
Keywords: Liver Fibrosis; Ultrasound Elastography; Shear wave speed; Stiffness; Liver Biopsy
MeSH Terms: conditions — Liver Cirrhosis; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 30 Patients with known liver biopsy results (Experimental): Patients with chronic liver disease with known biopsy results
  Interventions: Device: Sonographic SWE measurements with 4 different ultrasound systems

INTERVENTIONS:
Device: Sonographic SWE measurements with 4 different ultrasound systems — Sonographic Shear wave elastography will be performed to quantify liver fibrosis

SUMMARY:
Chronic liver disease is a major problem in the general population and there is an unmet need to diagnose(and screen) for liver disease with using noninvasive, cost-effective and sensitive techniques.The investigators hypothesize that variation using ultrasound elastography for the estimation of stage of liver fibrosis and steatosis in patients with diffuse liver disease exists due to different methods of measurements, and/or different systems. The proposed investigation is a cross-sectional study using ultrasound elastography and fat quantification modalities. The investigators are planning to enroll 30 subjects 18 years old and older in whom diffuse liver disease is suspected, and who have undergone non-focal liver biopsy in the past 6 months or are scheduled to undergo biopsy within 3 months of enrollment, as part of their routine clinical care. The investigators will use 4 different ultrasound devices with their shear wave elastography and speed of sound functions.

Specific aims;

* Compare shear wave elastography(SWE) measurements from different ultrasound systems; using histopathology as reference standards.
* Assess intra-operator and inter-operator reliability by measuring variability in elastography values by two operators on a single system.
* Determine the effect of deviations from guidelines(less number of measurements and measurements during active breath)

DETAILED DESCRIPTION:
Liver disease and cirrhosis are important causes of morbidity and mortality in the United States and are a major public health problem with 40,000 deaths and more than 1.4 billion dollars spent on medical services. Hepatic fibrosis is the final common pathway for many different liver insults and is known to be a dynamic process, which is reversible if diagnosed early and treated. If untreated, fibrosis eventually progresses to cirrhosis, which is irreversible. The diagnosis of fibrosis relies on liver biopsy (the gold standard) however, is an invasive procedure with risks and sampling errors. Indirect biomarkers of fibrogenesis can measure some of these components to determine categories of fibrosis, with a sensitivity and specificity of 47% and 90% respectively.It is shown in the literature that, fat content of liver is related with fibrosis development. Biopsy is accepted as the most accurate technique to assess liver fat and fibrosis amount.

Fibrotic livers demonstrate increased stiffness, a property that can be measured using technology named Ultrasound Elastography or sonoelastography (SWE). SWE is performed by insonating the patient with a low energy, amplitude, and frequency shear wave created by a vibrating probe. The propagated wave travels faster with increasing fibrosis: the stiffer the tissue, the faster the shear wave propagates. A pulse-echo ultrasound acquisition allows measurement of the wave velocity and the results are presented as kilopascals (kPa). Prior reports have described sensitivity and specificity for liver fibrosis detection of 80% and 97% respectively for SWE. The benefits of SWE are that it is inexpensive, reproducible, painless, rapid (< 10 min), easy to perform, and can be used for diagnosis, prognosis and monitoring disease progression.

The objective of this study is to compare the variation in elastography values and study the factors that might cause these variations.

The proposed investigation is a cross-sectional study using ultrasound elastography. The investigators are planning to enroll 30 subjects 18 years old and older in whom diffuse liver disease is suspected, and who have undergone non-focal liver biopsy in the past 6 months or are scheduled to undergo biopsy within 3 months of enrollment, as part of their routine clinical care.

All subjects will be required to come to the MGH main campus for 2 study visits within 60 days of each other. In addition, subjects will need to fast for at least 4 hours prior to study visits

There will be two visits in this study and maximum 60 days time frame between the visits is anticipated. Two operators will perform the ultrasound examination. Reproducibility and repeatability of the ultrasound devices will be estimated.

Ultrasound examination including sonoelastography will be performed using four FDA-approved ultrasound units; Both operators will perform;

* Median Elastograpy (10 measurements) on regular and variable map at a depth(in the area between 2cm from capsule and 6.5cm from skin)
* Median SWE value with active/free breath(10measurements)
* Median SWE value with less number of acquisitions(3measurements)

These measurements will be collected in subgroups using specific systems. In second visit, all measurements will be repeated with the same operators.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients
* Men or Woman
* Suspected diffuse liver disease and have had a liver biopsy within the last 6 months or are scheduled for a liver biopsy in the next 3 months.
* Consent to participate in the study

Exclusion Criteria:

* Pregnancy
* Acute illness/ cognitive impairment resulting in inability to cooperate with ultrasound
* Patients that do not consent to ultrasound examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony E. Samir, MD, MPH, Principal Investigator — Associate Medical Director, Ultrasound Imaging Services
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Younossi ZM, Stepanova M, Afendy M, Fang Y, Younossi Y, Mir H, Srishord M. Changes in the prevalence of the most common causes of chronic liver diseases in the United States from 1988 to 2008. Clin Gastroenterol Hepatol. 2011 Jun;9(6):524-530.e1; quiz e60. doi: 10.1016/j.cgh.2011.03.020. Epub 2011 Mar 25. PMID 21440669
- [Background] Mokdad AA, Lopez AD, Shahraz S, Lozano R, Mokdad AH, Stanaway J, Murray CJ, Naghavi M. Liver cirrhosis mortality in 187 countries between 1980 and 2010: a systematic analysis. BMC Med. 2014 Sep 18;12:145. doi: 10.1186/s12916-014-0145-y. PMID 25242656
- [Background] Pinzani M, Rombouts K. Liver fibrosis: from the bench to clinical targets. Dig Liver Dis. 2004 Apr;36(4):231-42. doi: 10.1016/j.dld.2004.01.003. PMID 15115333
- [Background] Scholmerich J, Holstege A. Aetiology and pathophysiology of chronic liver disorders. Drugs. 1990;40 Suppl 3:3-22. doi: 10.2165/00003495-199000403-00003. PMID 2081479
- [Background] Pellicoro A, Ramachandran P, Iredale JP, Fallowfield JA. Liver fibrosis and repair: immune regulation of wound healing in a solid organ. Nat Rev Immunol. 2014 Mar;14(3):181-94. doi: 10.1038/nri3623. PMID 24566915
- [Background] Actis GC, Olivero A, Lagget M, Pellicano R, Smedile A, Rizzetto M. The practice of percutaneous liver biopsy in a gastrohepatology day hospital: a retrospective study on 835 biopsies. Dig Dis Sci. 2007 Oct;52(10):2576-9. doi: 10.1007/s10620-006-9724-x. Epub 2007 Apr 12. PMID 17436094
- [Background] Cadranel JF, Rufat P, Degos F. Practices of liver biopsy in France: results of a prospective nationwide survey. For the Group of Epidemiology of the French Association for the Study of the Liver (AFEF). Hepatology. 2000 Sep;32(3):477-81. doi: 10.1053/jhep.2000.16602. PMID 10960438
- [Background] van der Poorten D, Kwok A, Lam T, Ridley L, Jones DB, Ngu MC, Lee AU. Twenty-year audit of percutaneous liver biopsy in a major Australian teaching hospital. Intern Med J. 2006 Nov;36(11):692-9. doi: 10.1111/j.1445-5994.2006.01216.x. PMID 17040353
- [Background] Sparchez Z. Complications after percutaneous liver biopsy in diffuse hepatopathies. Rom J Gastroenterol. 2005 Dec;14(4):379-84. PMID 16400355
- [Background] Bravo AA, Sheth SG, Chopra S. Liver biopsy. N Engl J Med. 2001 Feb 15;344(7):495-500. doi: 10.1056/NEJM200102153440706. No abstract available. PMID 11172192
- [Background] Rousselet MC, Michalak S, Dupre F, Croue A, Bedossa P, Saint-Andre JP, Cales P; Hepatitis Network 49. Sources of variability in histological scoring of chronic viral hepatitis. Hepatology. 2005 Feb;41(2):257-64. doi: 10.1002/hep.20535. PMID 15660389
- [Background] Regev A, Berho M, Jeffers LJ, Milikowski C, Molina EG, Pyrsopoulos NT, Feng ZZ, Reddy KR, Schiff ER. Sampling error and intraobserver variation in liver biopsy in patients with chronic HCV infection. Am J Gastroenterol. 2002 Oct;97(10):2614-8. doi: 10.1111/j.1572-0241.2002.06038.x. PMID 12385448
- [Background] Bedossa P, Dargere D, Paradis V. Sampling variability of liver fibrosis in chronic hepatitis C. Hepatology. 2003 Dec;38(6):1449-57. doi: 10.1016/j.hep.2003.09.022. PMID 14647056
- [Background] Friedrich-Rust M, Buggisch P, de Knegt RJ, Dries V, Shi Y, Matschenz K, Schneider MD, Herrmann E, Petersen J, Schulze F, Zeuzem S, Sarrazin C. Acoustic radiation force impulse imaging for non-invasive assessment of liver fibrosis in chronic hepatitis B. J Viral Hepat. 2013 Apr;20(4):240-7. doi: 10.1111/j.1365-2893.2012.01646.x. Epub 2012 Jul 31. PMID 23490368
- [Background] Fierbinteanu-Braticevici C, Andronescu D, Usvat R, Cretoiu D, Baicus C, Marinoschi G. Acoustic radiation force imaging sonoelastography for noninvasive staging of liver fibrosis. World J Gastroenterol. 2009 Nov 28;15(44):5525-32. doi: 10.3748/wjg.15.5525. PMID 19938190
- [Background] Ferraioli G, Tinelli C, Dal Bello B, Zicchetti M, Filice G, Filice C; Liver Fibrosis Study Group. Accuracy of real-time shear wave elastography for assessing liver fibrosis in chronic hepatitis C: a pilot study. Hepatology. 2012 Dec;56(6):2125-33. doi: 10.1002/hep.25936. Epub 2012 Aug 31. PMID 22767302
- [Background] Poynard T, Munteanu M, Luckina E, Perazzo H, Ngo Y, Royer L, Fedchuk L, Sattonnet F, Pais R, Lebray P, Rudler M, Thabut D, Ratziu V. Liver fibrosis evaluation using real-time shear wave elastography: applicability and diagnostic performance using methods without a gold standard. J Hepatol. 2013 May;58(5):928-35. doi: 10.1016/j.jhep.2012.12.021. Epub 2013 Jan 12. PMID 23321316
- [Background] Chen S, Sanchez W, Callstrom MR, Gorman B, Lewis JT, Sanderson SO, Greenleaf JF, Xie H, Shi Y, Pashley M, Shamdasani V, Lachman M, Metz S. Assessment of liver viscoelasticity by using shear waves induced by ultrasound radiation force. Radiology. 2013 Mar;266(3):964-70. doi: 10.1148/radiol.12120837. Epub 2012 Dec 6. PMID 23220900
- [Background] Goertz RS, Zopf Y, Jugl V, Heide R, Janson C, Strobel D, Bernatik T, Haendl T. Measurement of liver elasticity with acoustic radiation force impulse (ARFI) technology: an alternative noninvasive method for staging liver fibrosis in viral hepatitis. Ultraschall Med. 2010 Apr;31(2):151-5. doi: 10.1055/s-0029-1245244. Epub 2010 Mar 19. PMID 20306380
- [Background] Takahashi H, Ono N, Eguchi Y, Eguchi T, Kitajima Y, Kawaguchi Y, Nakashita S, Ozaki I, Mizuta T, Toda S, Kudo S, Miyoshi A, Miyazaki K, Fujimoto K. Evaluation of acoustic radiation force impulse elastography for fibrosis staging of chronic liver disease: a pilot study. Liver Int. 2010 Apr;30(4):538-45. doi: 10.1111/j.1478-3231.2009.02130.x. Epub 2009 Oct 27. PMID 19874490
- [Background] Friedrich-Rust M, Wunder K, Kriener S, Sotoudeh F, Richter S, Bojunga J, Herrmann E, Poynard T, Dietrich CF, Vermehren J, Zeuzem S, Sarrazin C. Liver fibrosis in viral hepatitis: noninvasive assessment with acoustic radiation force impulse imaging versus transient elastography. Radiology. 2009 Aug;252(2):595-604. doi: 10.1148/radiol.2523081928. PMID 19703889
- [Background] Wang QB, Zhu H, Liu HL, Zhang B. Performance of magnetic resonance elastography and diffusion-weighted imaging for the staging of hepatic fibrosis: A meta-analysis. Hepatology. 2012 Jul;56(1):239-47. doi: 10.1002/hep.25610. Epub 2012 Jun 6. PMID 22278368
- [Background] Sterling RK, Lissen E, Clumeck N, Sola R, Correa MC, Montaner J, S Sulkowski M, Torriani FJ, Dieterich DT, Thomas DL, Messinger D, Nelson M; APRICOT Clinical Investigators. Development of a simple noninvasive index to predict significant fibrosis in patients with HIV/HCV coinfection. Hepatology. 2006 Jun;43(6):1317-25. doi: 10.1002/hep.21178. PMID 16729309
- [Background] Cales P, Oberti F, Michalak S, Hubert-Fouchard I, Rousselet MC, Konate A, Gallois Y, Ternisien C, Chevailler A, Lunel F. A novel panel of blood markers to assess the degree of liver fibrosis. Hepatology. 2005 Dec;42(6):1373-81. doi: 10.1002/hep.20935. PMID 16317693
- [Background] Adams LA, Bulsara M, Rossi E, DeBoer B, Speers D, George J, Kench J, Farrell G, McCaughan GW, Jeffrey GP. Hepascore: an accurate validated predictor of liver fibrosis in chronic hepatitis C infection. Clin Chem. 2005 Oct;51(10):1867-73. doi: 10.1373/clinchem.2005.048389. Epub 2005 Jul 28. PMID 16055434
- [Background] Forns X, Ampurdanes S, Llovet JM, Aponte J, Quinto L, Martinez-Bauer E, Bruguera M, Sanchez-Tapias JM, Rodes J. Identification of chronic hepatitis C patients without hepatic fibrosis by a simple predictive model. Hepatology. 2002 Oct;36(4 Pt 1):986-92. doi: 10.1053/jhep.2002.36128. PMID 12297848
- [Background] Crespo G, Fernandez-Varo G, Marino Z, Casals G, Miquel R, Martinez SM, Gilabert R, Forns X, Jimenez W, Navasa M. ARFI, FibroScan, ELF, and their combinations in the assessment of liver fibrosis: a prospective study. J Hepatol. 2012 Aug;57(2):281-7. doi: 10.1016/j.jhep.2012.03.016. Epub 2012 Apr 17. PMID 22521355
- [Background] Rosenberg WM, Voelker M, Thiel R, Becka M, Burt A, Schuppan D, Hubscher S, Roskams T, Pinzani M, Arthur MJ; European Liver Fibrosis Group. Serum markers detect the presence of liver fibrosis: a cohort study. Gastroenterology. 2004 Dec;127(6):1704-13. doi: 10.1053/j.gastro.2004.08.052. PMID 15578508
- [Background] Wai CT, Greenson JK, Fontana RJ, Kalbfleisch JD, Marrero JA, Conjeevaram HS, Lok AS. A simple noninvasive index can predict both significant fibrosis and cirrhosis in patients with chronic hepatitis C. Hepatology. 2003 Aug;38(2):518-26. doi: 10.1053/jhep.2003.50346. PMID 12883497
- [Background] Imbert-Bismut F, Ratziu V, Pieroni L, Charlotte F, Benhamou Y, Poynard T; MULTIVIRC Group. Biochemical markers of liver fibrosis in patients with hepatitis C virus infection: a prospective study. Lancet. 2001 Apr 7;357(9262):1069-75. doi: 10.1016/S0140-6736(00)04258-6. PMID 11297957

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All 30 patients were scanned in clinic ultrasound setting. 2 visits were scheduled for each patient. Mean difference between visits was 11 days. Mean difference between liver biopsy date and first visit date was 89 days. 2 patients were lost to followup for 2nd visit.
Groups:
- Chronic Liver Disease Patients With Known Liver Biopsy Results: Patients with chronic liver disease with known biopsy results
  Sonographic SWE measurements with Toshiba/Canon APLIO500: Sonographic Shear wave elastography will be performed to quantify liver fibrosis
  Sonographic SWE measurements with Siemens ACUSON S3000: Sonographic Shear wave elastography will be performed to quantify liver fibrosis
  Sonographic SWE measurements with GE LOGIQ E9: Sonographic Shear wave elastography will be performed to quantify liver fibrosis
  SWE measurements with FibroScan: Transient elastography will be performed to quantify liver fibrosis
Period: Overall Study
Arm/Group | Chronic Liver Disease Patients With Known Liver Biopsy Results
Started | 30
Completed | 28
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- 30 Patients With Known Liver Biopsy Results: Patients with chronic liver disease with known biopsy results
  Sonographic SWE measurements with Toshiba APLIO500: Sonographic Shear wave elastography will be performed to quantify liver fibrosis
  Sonographic SWE measurements with Siemens ACUSON S3000: Sonographic Shear wave elastography will be performed to quantify liver fibrosis
  Sonographic SWE measurements with GE LOGIQ E9: Sonographic Shear wave elastography will be performed to quantify liver fibrosis
  SWE measurements with FibroScan: Transient elastography will be performed to quantify liver fibrosis
  Sonographic speed of sound measurements with GE LOGIQ E9: Sonographic speed of sound function of the machine will be used to quantify liver steatosis
Arm/Group | 30 Patients With Known Liver Biopsy Results
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 49 [21 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Fibrosis stage [Number; unit: participants] — Fibrosis severity in the biopsy samples were staged using METAVIR system. Higher stages correspond to higher disease severity, and stage4 shows cirrhosis.
  participants
    Fibrosis 0 | 10
    Fibrosis 1 | 7
    Fibrosis 2 | 3
    Fibrosis 3 | 5
    Fibrosis 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Deviations From Suggested Guidelines- Any Effect on Agreement
Description: We collected guideline suggested shear wave elastography measurements from 20 patients. Guidelines suggest collecting 1) 10 measurements, 2) Asking patient to hold breath during the measurements. As a deviation from guideline suggestions, we collected measurements during free breath movements without asking patient to hold breath. As a deviation from the guideline suggestions, fewer number of measurements (3 measurements) were collected with asking the patient to hold breath during the measurements. All measurements were collected using one type of ultrasound system. All measurements were collected by 2 operators in 2 visits.
Time Frame: Visit 1 and Visit 2, an average of 2.5 hours for each visit
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Groups:
- Guideline Suggested Measurements: 10 measurements in an area between 2cm from liver capsule and 6.5cm from skin
- Fewer Number of Measurements: 3 SWE measurements were collected.
- Free Breath Measurements: 10 SWE measurements were collected during free breath
Arm/Group | Guideline Suggested Measurements | Fewer Number of Measurements | Free Breath Measurements
Number analyzed (Participants) | 20 | 20 | 20
correlation coefficient
  ICC for inter-operator agreement in visit1 | 0.77 [0.45 to 0.90] | 0.75 [0.40 to 0.90] | 0.69 [0.26 to 0.87]
  ICC for inter-operator agreement in visit2 | 0.86 [0.64 to 0.94] | 0.80 [0.48 to 0.92] | 0.68 [0.20 to 0.87]
  ICCfor intra-op agreement between 2 visits for op1 | 0.94 [0.84 to 0.97] | 0.90 [0.75 to 0.96] | 0.93 [0.61 to 0.98]
  ICCfor intra-op agreement between 2 visits for op2 | 0.89 [0.74 to 0.96] | 0.89 [0.73 to 0.96] | 0.95 [0.87 to 0.98]

2. Primary Outcome: Interoperator and Intraoperator Agreement in m/s and kPA Units
Description: In 20 patients we collected 10 shear wave elastography measurements in m/s and kPA units. Using one of the available ultrasound systems, 2 operators collected these measurements in 2 visits. Theoretically, m/s to kPA conversion can be made using an equation. However, some systems provide opportunity to get data in both units. Although algebraically m/s and kPA can be converted to each other, we found some minor differences in terms of inter-operator and intra-operator agreement.
Time Frame: Visit 1 and Visit 2, an average of 2.5 hours for each visit
Measure: Number (95% Confidence Interval); unit: Intraclass correlation coefficient value
Groups:
- Measurements in m/s Unit; Measurements in kPA Unit: In 20 patients, we collected 10 measurements at a depth between 2cm from liver capsule and 6.5 from skin.
Arm/Group | Measurements in m/s Unit | Measurements in kPA Unit
Number analyzed (Participants) | 20 | 20
Intraclass correlation coefficient value
  ICC for inter-operator agreement in visit1 | 0.87 [0.47 to 0.96] | 0.84 [0.36 to 0.95]
  ICC for inter-operator agreement in visit2 | 0.80 [0.26 to 0.94] | 0.77 [0.13 to 0.94]
  ICC for intra-operator agreement for opt1 | 0.92 [0.71 to 0.97] | 0.88 [0.57 to 0.96]
  ICC for intra-operator agreement for opt2 | 0.81 [0.35 to 0.94] | 0.78 [0.27 to 0.94]

ADVERSE EVENTS:
Time Frame: Adverse events were not expected for this study. 0 participants were at risk for this study. Adverse events were not collected.
Description: We used ultrasound systems and ultrasound is a very safe technique for liver evaluation. There are no expected risks for this technique. Therefore, all-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed. 0 participants were at risk for this study.
Arm/Group | 30 Patients With Known Liver Biopsy Results
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
* Reference standard (biopsy) was collected from medical records. Pathology slides were not re-evaluated.
* Low number of patients to perform diagnostic performance analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT03342560/Prot_SAP_000.pdf